CLINICAL TRIAL: NCT00790192
Title: A Phase 3 Randomized, Double-Blind, Placebo- and Active Comparator-Controlled Clinical Trial to Study the Efficacy and Safety of Two Doses of Lurasidone in Acutely Psychotic Subjects With Schizophrenia (PEARL 3)
Brief Title: Lurasidone HCL - A 6-week Phase 3 Study of Patients With Acute Schizophrenia.
Acronym: PEARL 3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D1050233
Record Dates: First submitted 2008-11-10; First posted 2008-11-13 (Estimated); Results first posted 2011-10-06 (Estimated); Last update posted 2016-03-17 (Estimated); Status verified 2016-03

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; SM-13496; Latuda; Lurasidone
MeSH Terms: conditions — Schizophrenia | interventions — Lurasidone Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Lurasidone 80mg (Experimental)
  Interventions: Drug: Lurasidone
- Lurasidone 160mg (Experimental)
  Interventions: Drug: Lurasidone
- Quetiapine XR (Active Comparator)
  Interventions: Drug: Quetiapine XR
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lurasidone — Lurasidone 80 mg tablets
  Arms: Lurasidone 80mg
Drug: Lurasidone — Lurasidone 4 40 mg tablets
  Arms: Lurasidone 160mg
Drug: Quetiapine XR — Quetiapine XR 600mg
  Arms: Quetiapine XR
Drug: Placebo — Matching Placebo to Lurasidone or Quetiapine
  Arms: Placebo

SUMMARY:
Lurasidone HCl is a compound being developed for the treatment of schizophrenia. This clinical study is designed to test the hypothesis that lurasidone is effective, tolerable, and safe as compared with quetiapine XR short term among acutely psychotic patients with chronic schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent and aged between 18 and 75 years of age.
* Meets DSM-IV™ criteria for a primary diagnosis of schizophrenia.
* Not pregnant, if of reproductive potential agrees to remain abstinent or use adequate and reliable contraception for duration of study.
* Able and agrees to remain off prior antipsychotic medication for the duration of study.
* Good physical health on the basis of medical history, physical examination, and laboratory screening.
* Willing and able to comply with the protocol, including the inpatient requirements and outpatient visits.

Exclusion Criteria:

* Considered by the investigator to be at imminent risk of suicide or injury to self, others, or property.
* Any chronic organic disease of the CNS (other than schizophrenia).
* Used investigational compound within 30 days.
* Clinically significant or history of alcohol abuse/alcoholism or drug abuse/dependence within the last 6 months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 488 (Actual)
Dates: Start 2008-10; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, MD, Study Director — Sumitomo Pharma America, Inc.
Locations (65):
- United States (29):
  - K&S Professional Research Services, LLC, Little Rock, Arkansas
  - Woodland International Research Group, Little Rock, Arkansas
  - Clinical Pharmacological Studies, Inc., Cerritos, California
  - Comprehensive Neuroscience, Inc, Cerritos, California
  - Clinical Innovations, Inc., Costa Mesa, California
  - Synergy Escondido, Escondido, California
  - Collaborative Neuroscience Network, Garden Grove, California
  - Apostle Clinical Trials, Inc., Long Beach, California
  - California Clinical Trials, Paramount, California
  - Pasadena Research Institute, Pasadena, California
  - CNRI-Los Angeles. LLC, Pico Rivera, California
  - Clinical Innovations, Inc., Riverside, California
  - CNRI-San Diego, San Diego, California
  - UCSD Medical Center, Sandeigo, California
  - Segal Institute for Clinical Research, Highlands Ranch, Colorado
  - Comprehensive Neuroscience, Inc., Washington D.C., District of Columbia
  - Florida Clinical Research Center, Bradenton, Florida
  - Florida Clinical Research Center, LLC, Fruitland Park, Florida
  - Lake Charles Clinical Trials, Lake Charles, Louisiana
  - Booker, J. Gary, MD. APMC, Shreveport, Louisiana
  - Precise Clinical Research, Flowood, Mississippi
  - St. Charles Psychiatric Associates, Saint Charles, Missouri
  - St. Louis Research, Inc., St Louis, Missouri
  - CRI Worldwide, Willingboro, New Jersey
  - Comprehensive Neuroscience, Inc, Holliswood, New York
  - Segal Institute for Clinical Research, Winston-Salem, North Carolina
  - Community Clinical Research, Austin, Texas
  - Future Search Trials of Neurology, Austin, Texas
  - Pillar Clinical Research, Dallas, Texas
- India (10):
  - S.V. Medical College, Tirupati, Andhra Pradesh
  - Vijayawada Institute of Mental Health and Neurosciences, Vijayawada, Andhra Pradesh
  - Seth K M School of P G Medicine & Research, Ahmedabad, Gujarat
  - SBKS Medical Institute and Research Centre, Vadodara, Gujarat
  - Justice K.S. Hegde Charitable Hospital, Mangalore, Karnataka
  - JSS Medical College and Hospital, Mysore, Karnataka
  - Shanti Nursing Home, Aurangabad, Maharashtra
  - Deenanath Mangeshkar Hospital and Research Centre, Pune, Maharashtra
  - Mahatma Gandhi Institute of Medical Sciences, Sewāgrām, Maharashtra
  - Madras Medical College & Government General Hospital, Chennai, Tamil Nadu
- Romania (6):
  - Spitalul Clinic Judetean de Urgenta Arad, Str. Octavian Goga Nr. 17, Arad
  - Spitalul de Psihiatrie Titan "Dr. Constantin Gorgos", Bdul Nicolae Grigorescu Nr. 41, București
  - Spitalul Clinic de Psihiatrie Prof. Dr. Alexandru Obregia, Sos. Berceni Nr. 10-12, București
  - Spitalul Judetean Arges, Str. Negru Voda Nr. 53, Pitesti
  - Spitalul Clinic de Psihiatrie Prof. Dr. Alexandru Obregia, Bucharest
  - Spitalul Clinic de Neurologie si Psihiatrie Oradea, Oradea
- Russia (11):
  - SEI of H.P. Educat. Northern SMU, Arkhangelsk
  - St. Petersburg SHI Psychiatrical Hosptial #1 n.a. Kaschenko, Gatchina
  - Moscow Scientific Research Institute of Psychiatry, Moscow
  - Institution of RAMS Mental Health Research Center of RAMS, Moscow
  - City Clinical Psichiatric Hospital #1, Nizhny Novgorod
  - City Psychiatric Hospital #2 of St. Nikolay Chudotvorets, Saint Petersburg
  - City Psychiatric Hospital #3 of Skvortsov-Stepanov, Saint Petersburg
  - City Psychiatric Hospital #4, Saint Petersburg
  - SHI City Psychoneurological Dispensary #7, Saint Petersburg
  - St. Petersburg GUZ City Psychiatric Hospital #6, Saint Petersburg
  - SHI Samara Psychiatric Hospital, Samara
- Ukraine (9):
  - Kherson Regional Psychiatric Hospital, Kherson,vil., Stepanovka
  - RCH n.a.I.I.Mechnikov, Reg.Cent. of Psychosom. Pathology, Dnipropetrovsk
  - Chair of Psychiatry and Medical Psychology, Donetsk
  - Centre of Novel Treatment and Rehabilitation of Psychotic disorders, Kyiv
  - Kyiv City Psychoneurological Hospital, Kyviv
  - Lviv Reg.St.Cl.Psych.Hosp, Lviv
  - Reg. Psychiatric Hospital, Odesa
  - Poltava Regional Clinical Psychiatric Hospital,, Poltava
  - Crimean republican Clinical Psychiatric Hospital, Simferopol

REFERENCES:
- [Result] Loebel A, Cucchiaro J, Sarma K, Xu L, Hsu C, Kalali AH, Pikalov A, Potkin SG. Efficacy and safety of lurasidone 80 mg/day and 160 mg/day in the treatment of schizophrenia: a randomized, double-blind, placebo- and active-controlled trial. Schizophr Res. 2013 Apr;145(1-3):101-9. doi: 10.1016/j.schres.2013.01.009. Epub 2013 Feb 13. PMID 23415311
- [Result] Harvey PD, Siu CO, Hsu J, Cucchiaro J, Maruff P, Loebel A. Effect of lurasidone on neurocognitive performance in patients with schizophrenia: a short-term placebo- and active-controlled study followed by a 6-month double-blind extension. Eur Neuropsychopharmacol. 2013 Nov;23(11):1373-82. doi: 10.1016/j.euroneuro.2013.08.003. Epub 2013 Aug 27. PMID 24035633
- [Result] Loebel AD, Siu CO, Cucchiaro JB, Pikalov AA, Harvey PD. Daytime sleepiness associated with lurasidone and quetiapine XR: results from a randomized double-blind, placebo-controlled trial in patients with schizophrenia. CNS Spectr. 2014 Apr;19(2):197-205. doi: 10.1017/S1092852913000904. Epub 2013 Dec 13. PMID 24330860
- [Derived] Hopkins SC, Tomioka S, Ogirala A, Loebel A, Koblan KS, Marder SR. Assessment of Negative Symptoms in Clinical Trials of Acute Schizophrenia: Test of a Novel Enrichment Strategy. Schizophr Bull Open. 2022 Apr 7;3(1):sgac027. doi: 10.1093/schizbullopen/sgac027. eCollection 2022 Jan. PMID 39144777
- [Derived] Hopkins SC, Ogirala A, Worden M, Koblan KS. Depicting Safety Profile of TAAR1 Agonist Ulotaront Relative to Reactions Anticipated for a Dopamine D2-Based Pharmacological Class in FAERS. Clin Drug Investig. 2021 Dec;41(12):1067-1073. doi: 10.1007/s40261-021-01094-7. Epub 2021 Nov 9. PMID 34751928
- [Derived] Harvey PD, Siu CO, Ogasa M, Loebel A. Effect of lurasidone dose on cognition in patients with schizophrenia: post-hoc analysis of a long-term, double-blind continuation study. Schizophr Res. 2015 Aug;166(1-3):334-8. doi: 10.1016/j.schres.2015.06.008. Epub 2015 Jun 24. PMID 26117157
- [Derived] Nasrallah HA, Cucchiaro JB, Mao Y, Pikalov AA, Loebel AD. Lurasidone for the treatment of depressive symptoms in schizophrenia: analysis of 4 pooled, 6-week, placebo-controlled studies. CNS Spectr. 2015 Apr;20(2):140-7. doi: 10.1017/S1092852914000285. Epub 2014 Jun 23. PMID 24955752

RESULTS

PARTICIPANT FLOW:
Groups:
- Lurasidone 80 mg: Lurasidone 80 mg tablets taken orally once a day
- Lurasidone 160 mg: Lurasidone 160 mg (4 tablets) taken orally once a day
- Quetiapine XR 600mg: Quetiapine XR 600 mg (4 tablets) orally taken once a day
- Placebo: Matching placebo to either lurasidone or quetiapine XR. The total for this group is 73 and the adverse events only add up to 69 because the total is based on all treatment emergent adverse events not limited to >= 5%.
Period: Overall Study
Arm/Group | Lurasidone 80 mg | Lurasidone 160 mg | Quetiapine XR 600mg | Placebo
Started | 125 | 121 | 120 | 122
Completed | 89 | 93 | 97 | 74
Not Completed | 36 | 28 | 23 | 48

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lurasidone 80 mg | Lurasidone 160 mg | Quetiapine XR 600mg | Placebo | Total
Number analyzed (Participants) | 125 | 121 | 120 | 122 | 488
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.2 (10.9) | 37.9 (11.3) | 37.4 (10.4) | 37.4 (10.8) | 37.2 (10.8)
Gender [Number; unit: participants] — There were two subjects, one randomized to the Quetiapine 600 mg group and one subject randomized to placebo that did not take study drug. Thus you see a discrepancy between the participant population and the overall baseline population for the two treatment groups (1 less patient in each treatment arm).
  participants
    Female | 29 | 39 | 42 | 44 | 154
    Male | 96 | 82 | 77 | 77 | 332
Region of Enrollment [Number; unit: participants] — There were two subjects, one randomized to the Quetiapine 600 mg group and one subject randomized to placebo that did not take study drug. Thus you see a discrepancy between the participant population and the overall baseline population(1 less patient in each treatment arm).
  participants
    United States | 40 | 37 | 35 | 39 | 151
    Ukraine | 19 | 20 | 19 | 17 | 75
    Romania | 13 | 11 | 13 | 12 | 49
    Russian Federation | 22 | 22 | 21 | 22 | 87
    India | 24 | 25 | 25 | 24 | 98
    Colombia | 7 | 6 | 6 | 7 | 26

OUTCOME MEASURES:

1. Primary Outcome: Primary Efficacy Endpoint: Mean Change in Total PANSS Score From Baseline to the End of the Double Blind Phase
Description: The PANSS (Positive and Negative Syndrome Scale) is a 30-item scale (range 30-210) designed to assess various symptoms of schizophrenia including delusions, grandiosity, blunted affect, poor attention, and poor impulse control. The 30 symptoms are rated on a 7-point scale that ranges from 1 (absent) to 7 (extreme psychopathology). The PANSS total score consists of the sum of all 30 PANSS items. Higher scores indicate worsening.
Time Frame: Week 6
Population: The primary population for the efficacy analysis was the Intent-to-Treat (ITT) population. All subjects who were randomized, received at least one dose of study medication, and have a Baseline efficacy measurement and at least one post-Baseline efficacy measurement, were in the efficacy analysis in the treatment group to which they were randomized.
Measure: Least Squares Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | Lurasidone 80 mg | Lurasidone 160 mg | Quetiapine XR 600mg | Placebo
Number analyzed (Participants) | 125 | 121 | 116 | 120
scores on a scale | -22.2 [-25.7 to -18.7] | -26.5 [-30.0 to -23.0] | -27.8 [-31.3 to -24.2] | -10.3 [-13.9 to -6.7]
Statistical Analysis 1: Comparison: Lurasidone 80 mg vs Lurasidone 160 mg vs Quetiapine XR 600mg vs Placebo; Test type: Superiority or Other; p < 0.05, Mixed Models Analysis

2. Secondary Outcome: Secondary Outcome: CGI-S From Baseline to the End of the Double-blind Treatment
Description: Clinical Global Impression of Severity is a clinician-rated assessment of the subject's current illness state on a 7 point scale, where a higher score is associated with greater illness severity. The scale has a single item measured on a 7 point scale from 1 ('normal', not ill) to 7 (extremely ill).
Time Frame: 6-Weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | Lurasidone 80 mg | Lurasidone 160 mg | Quetiapine XR 600mg | Placebo
Number analyzed (Participants) | 125 | 121 | 116 | 120
scores on a scale | -1.5 [-1.7 to -1.3] | -1.7 [-1.9 to -1.5] | -1.7 [-1.9 to -1.5] | -0.9 [-1.1 to -0.7]
Statistical Analysis 1: Comparison: Lurasidone 80 mg vs Lurasidone 160 mg vs Quetiapine XR 600mg vs Placebo; Test type: Superiority or Other; p < 0.05, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: 14 days post study therapy
Arm/Group | Lurasidone 80 mg | Lurasidone 160 mg | Quetiapine XR 600mg | Placebo
Serious Adverse Events (participants affected / at risk) | 1/125 | 4/121 | 1/119 | 4/121
Other Adverse Events (participants affected / at risk) | 71/125 | 76/121 | 70/119 | 69/121
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lurasidone 80 mg (N=125) | Lurasidone 160 mg (N=121) | Quetiapine XR 600mg (N=119) | Placebo (N=121)
Left Ventricular Dysfunction (Cardiac disorders) | 1 (1) | 4 (4) | 1 (1) | 4 (4)
Abdominal Hernia Obstructive (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac Chest Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatitis Viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (119) | 0 (0)
Hand Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Agression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyschotic Disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Schizophrenia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Suicidal Behavior (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Suicidal Ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Physical Assault (Social circumstances) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Labile Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lurasidone 80 mg (N=125) | Lurasidone 160 mg (N=121) | Quetiapine XR 600mg (N=119) | Placebo (N=121)
Constipation (Gastrointestinal disorders) | 3 (3) | 1 (1) | 8 (8) | 3 (3)
Dry Mouth (Gastrointestinal disorders) | 2 (2) | 2 (2) | 9 (9) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 3 (3) | 7 (7) | 3 (3) | 4 (4)
Nausea (Gastrointestinal disorders) | 10 (10) | 8 (8) | 4 (4) | 4 (4)
Vomiting (Gastrointestinal disorders) | 8 (8) | 9 (9) | 6 (6) | 6 (6)
Upper Respiratory Tract Infection (Infections and infestations) | 2 (2) | 1 (1) | 6 (6) | 1 (1)
Weight Increase (Investigations) | 1 (1) | 2 (2) | 8 (8) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 7 (7) | 1 (1)
Akathisia (Nervous system disorders) | 10 (10) | 9 (9) | 2 (2) | 1 (1)
Dizziness (Nervous system disorders) | 6 (6) | 7 (7) | 16 (16) | 2 (2)
Headache (Nervous system disorders) | 12 (12) | 12 (12) | 13 (13) | 13 (13)
Parkinsonism (Nervous system disorders) | 7 (7) | 8 (8) | 4 (4) | 0 (0)
Somnolence (Nervous system disorders) | 5 (5) | 8 (8) | 16 (16) | 1 (1)
Agitation (Psychiatric disorders) | 4 (4) | 6 (6) | 3 (3) | 10 (10)
Anxiety (Psychiatric disorders) | 9 (9) | 4 (4) | 1 (1) | 10 (10)
Insomnia (Psychiatric disorders) | 14 (14) | 8 (8) | 5 (5) | 11 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No